CLINICAL TRIAL: NCT04501822
Title: One-year Cardiac Follow-up of Patients With COVID-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: TCRC-COVID
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Cardiac Complication
Keywords: Covid19; Cardiovascular Disease; Echocardiography
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19 pneumonia patients: The study includes men and women ≥18 years old with documented COVID-19 pneumonia
  Interventions: Diagnostic Test: Evaluation of clinical, instrumental and laboratory diagnostics tests

INTERVENTIONS:
Diagnostic Test: Evaluation of clinical, instrumental and laboratory diagnostics tests — During follow-up visits patients undergo clinical, instrumental and laboratory diagnostics tests

SUMMARY:
The primary objective of the study is to assess the cardiac status of COVID-19 pneumonia patients during 1 year after discharge

DETAILED DESCRIPTION:
Although COVID-19 manifests in most cases with respiratory symptoms, cardiovascular abnormalities is common in hospitalized patients. Patients with cardiovascular risk factors or established disease appear to have a worse prognosis. Myocardial dysfunction could be a direct manifestation of COVID-19. The investigators hypothesize that subjects after COVID-19 pneumonia present myocardial and vascular remodeling during 1 year after discharge, even in the absence of prior cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

-Patients with documented COVID-19 pneumonia

Exclusion Criteria:

* Patients with cancer
* Impossible to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes men and women ≥18 years old with documented COVID-19 pneumonia
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2020-07-19 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Echocardiographic assessment of cardiac function | up to one year
  Echocardiographic assessment of global strain parameters at 3 and 12 months after discharge

SECONDARY OUTCOMES:
МАССЕ | up to one year
  Major adverse cardiac and cerebrovascular events: cardiac death, myocardial infarction, or stroke at 3 and 12 months after discharge
Quantitative analysis of parenchymal lung damage | up to one year
  Describe the parenchymal lung damage through a quantitative analysis with chest CT at 3 and 12 months after discharge
Functional exercises capacity assessment | up to one year
  Six-min walk test at 3 and 12 months after discharge
Evaluation of renal function | up to one year
  Measure of creatinine clearance at 3 and 12 months after discharge
Evaluation of inflammation | up to one year
  Analysis for C-reactive protein at 3 and 12 months after discharge
Evaluation of coagulation abnormality | up to one year
  Analysis for activated clotting time at 3 and 12 months
Evaluation of quality of life in first year after discharge | up to one year
  Assessment of the Short Form Health Survey (SF36) at 3 and 12 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Elena Yaroslavskaya, PhD, Principal Investigator — Tyumen Cardiology Research Center
Locations (1):
- Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tyumen, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT04501822/Prot_000.pdf